CLINICAL TRIAL: NCT04478136
Title: Can Blood Panels Provide Early Warning of Bleeding in Patients on ECMO?
Status: Withdrawn | Type: Observational
Why Stopped: This protocol was never initiated
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-10472
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: ECMO; Bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Major bleeders (MB): Additional blood to be drawn from patients on ECMO who have a major bleeding event.
  Interventions: Diagnostic Test: Blood test of factor levels
- Non-major bleeders (NMB)

INTERVENTIONS:
Diagnostic Test: Blood test of factor levels — Blood draw from central line to check coagulation factors
  Groups: Major bleeders (MB)

SUMMARY:
This is a prospective, observational study of 60 adult patients anticoagulated with bivalirudin for extracorporeal membrane oxygenation (ECMO). The study aims to identify the most precise early warning blood test or panel of blood tests to predict bleeding in patients on bivalirudin/ECMO. The project will involve comparing currently used blood tests with an extended panel of coagulation and metabolic blood tests with the aim of early warning of impending bleeding to allow intervention in the form of adjusted bivalirudin dose, modification of other risk factors, or transfusion with hemostatic products targeted to documented coagulation test abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 - 70 years who are anticoagulation (AC) with bivalirudin and placed on ECMO for cardiac and/or respiratory failure. Surgical and non-surgical patients will be included.

Exclusion Criteria:

* known pre-existing bleeding disorder (due to a factor deficiency that requires factor replacement, or platelet disorder), or a creatinine > 2.0.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population in this prospective cohort study will include sixty (60) adults 18 - 70 years who are anticoagulation (AC) with bivalirudin and placed on ECMO for cardiac and/or respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with changes in extended blood panel (EBP) for each of the bleeding and non-bleeding patient groups. | Up to 2 weeks
  To determine if changes over time in an extended blood panel (EBP) and metabolic panel (MP) could provide early warning of impending bleeding in patients on ECMO.
  The extended blood panel includes: Dilute thrombin time (DTT), Factor XIII, Factor VIII, Factor IX, and Von Willebrand Disease (VWD) panel, and Factor XI, Factor X, Factor VII, Factor V, Factor II, protein C, protein S, thromboelastogram (TEG), and TEG-platelet mapping).

SECONDARY OUTCOMES:
Number of participants designated as major bleeders (MB) | Up to 2 weeks
Number of participants designated as non-major bleeders (NMB) | Up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kiri Mackersey, MBChB, Principal Investigator — Albert Einstein College

IPD SHARING:
Plan to Share IPD: No